CLINICAL TRIAL: NCT05083377
Title: Clozapine Use Pattern in the Province of Seville
Status: Completed | Type: Observational
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Sponsor
Other Study IDs: CLOZASEV
Record Dates: First submitted 2021-10-06; First posted 2021-10-19 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Schizophrenia and Related Disorders
Keywords: clozapine
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who have been prescribed clozapine during 2018: Patients who have been prescribed (initially or regularly) clozapine during 2018, based on the casuistry provided by the Pharmacy service of the different hospitals.

SUMMARY:
CLOZAPINE USE PATTERN IN THE PROVINCE OF SEVILLE

DETAILED DESCRIPTION:
Subjects with a diagnosis of schizophrenia (F20 of ICD-10) under treatment with clozapine in the province of Seville. The use of clozapine, variability between centers and treatment modification will be identified.

ELIGIBILITY:
Inclusion Criteria:

Patients who have been prescribed (initially or regularly) clozapine during 2018, based on the casuistry provided by the Pharmacy service of the different hospitals.

Exclusion Criteria:

* Parkinson's disease
* Dementia

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have been prescribed (initially or regularly) clozapine during 2018, based on the casuistry provided by the Pharmacy service of the different hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2020-09-08 (Actual); Primary Completion 2021-09-08 (Actual); Study Completion 2021-09-08 (Actual)

PRIMARY OUTCOMES:
Identify the pattern of clozapine use in the province of Seville | year 2018
  Identify the pattern of clozapine use in the province of Seville

SECONDARY OUTCOMES:
Analyze the variability between centers or professionals | year 2018
  Analyze the variability between centers or professionals
Analyze the changes in the course of the disease since the prescription of clozapine | year 2018
  Analyze the changes in the course of the disease since the prescription of clozapine

CONTACTS AND LOCATIONS:
Overall Officials: Benedicto Crespo Facorro, Professor, Principal Investigator — benedicto.crespo.sspa@juntadeandalucia.es
Locations (1):
- Hospital Universitario Virgen del Rocío, Seville, Spain